CLINICAL TRIAL: NCT02770417
Title: Oral β-Alanine Supplementation in Patients With COPD: Structural, Metabolic and Functional Adaptations
Brief Title: Oral β-Alanine Supplementation in Patients With COPD
Acronym: BACOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Martijn Spruit, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BACOPD
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- COPD (beta-alanine) (Active Comparator)
  Interventions: Dietary Supplement: beta-alanine
- COPD (placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- Healthy controls (Other)
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: beta-alanine — Patients receive beta-alanine
  Arms: COPD (beta-alanine)
Dietary Supplement: placebo — Patients receive placebo
  Arms: COPD (placebo)
Other: control — Healthy controls will be assessed to compare baseline muscle carnosine levels
  Arms: Healthy controls

SUMMARY:
Preliminary evidence suggest that patients with chronic obstructive pulmonary disease (COPD) suffer from lower-limb muscle dysfunction. This may, at least in part, be due to a combination of physical inactivity and muscle oxidative stress. Pilot data (not published) clearly show that patients with COPD have significantly lower carnosine, which is a pH (acidity-basicity level) buffer and antioxidant, levels in the m. vastus lateralis compared to healthy subjects. Beta-alanine supplementation has shown to increase muscle carnosine in trained and untrained healthy subjects. This study will assess if muscle carnosine can be augmented by beta-alanine supplementation in 40 COPD patients (20 patients receive beta-alanine, 20 patients receive placebo). 10 healthy elderly controls will also be assessed to compare baseline muscle carnosine levels.

The aims of this study are to:

1. Investigate baseline muscle carnosine levels to confirm the pilot data in a larger sample of patients with COPD compared with healthy elderly subjects
2. Investigate if beta-alanine supplementation augments muscle carnosine in COPD patients and whether it has an influence on exercise capacity, lower-limb muscle function and quality of life
3. To investigate baseline and post supplementation structural and metabolic muscle characteristics and markers of oxidative stress and inflammation in COPD patients and it's association with muscle carnosine levels

ELIGIBILITY:
Inclusion Criteria:

* COPD: diagnosis of moderate to very severe COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
* Healthy controls: forced expiratory volume at one second/forced vital capacity (FEV1/FVC) > 0.7, matched for age and gender

Exclusion Criteria:

* The presence of known instable cardiac disease
* neurological disease and/or musculoskeletal disease that preclude safe participation in an exercise test
* a history of drugs/alcohol abuse
* vegetarianism
* inability to understand the Flemish language.

COPD-specific exclusion criteria:

* COPD exacerbation and/or hospitalization in the last 6 weeks
* participation in pulmonary rehabilitation in the previous 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
muscle carnosine | change from baseline to 12 weeks
  by means of high pressure liquid chromatography(HPLC)-analysis of a muscle biopsy
maximal exercise capacity | change from baseline to 12 weeks
  by means of an incremental maximal cycle test
submaximal exercise capacity | change from baseline to 12 weeks
  by means of a constant-work rate cycle test

SECONDARY OUTCOMES:
Functional exercise test 1 | change from baseline to 12 weeks
  by means of a 6 minutes walk test
Functional exercise test 2 | change from baseline to 12 weeks
  by means of a 4 meter gait test
Muscle function quadriceps | change from baseline to 12 weeks
  by means of measuring quadriceps (isometric and isokinetic knee extension-flexion)
Respiratory muscle function | change from baseline to 12 weeks
  by means of measuring respiratory muscle strength (maximal inspiratory and expiratory pressure)
Muscle function hand grip | change from baseline to 12 weeks
  by means of measuring hand grip strength
Muscle characteristics | change from baseline to 12 weeks
  Structural and metabolic parameters will be measured with dedicated methodology
Blood parameters submaximal exercise test | change from baseline to 12 weeks
  by means of obtaining venous blood before, during and after the constant-work rate cycle test. Blood parameters will be measured with dedicated methodology.
Blood parameters fasted state | change from baseline to 12 weeks
  by means of obtaining fasting venous blood. Blood parameters will be measured with dedicated methodology.
Blood parameters maximal exercise test | change from baseline to 12 weeks
  by means of obtaining venous blood before and after the maximal cycle test. Blood parameters will be measured with dedicated methodology.
Comorbidities | change from baseline to 12 weeks
  by means of Charlson Morbidity index
Comorbidities: ankle-brachial pressure index | change from baseline to 12 weeks
  by means of ankle-brachial pressure index
Comorbidities blood pressure | change from baseline to 12 weeks
  by means of resting systolic and diastolic blood pressure
Comorbidities body composition 1 | change from baseline to 12 weeks
  by means of bio-electrical impedance
Comorbidities body composition 2 | change from baseline to 12 weeks
  by means of whole body dual X-ray absorptiometry
Quality of life: anxiety and depression | change from baseline to 12 weeks
  by means of the "Hospital Anxiety and Depression Scale"
Quality of life: fatigue | change from baseline to 12 weeks
  by means of the "Multidimensional Fatigue Inventory"
Quality of life: dyspnea | change from baseline to 12 weeks
  by means of the " Modified Medical Research Council (MMRC) dyspnea grade"
Quality of life: general | change from baseline to 12 weeks
  by means of the "Euroqol 5 dimensions (EQ-5D) generic questionnaire"
Quality of life: COPD | change from baseline to 12 weeks
  by means of the "COPD assessment test"
Physical activity: accelerometer | change from baseline to 12 weeks
  by means of physical activity monitoring via Actigraph (accelerometer)
Physical activity: questionnaire 1 | change from baseline to 12 weeks
  by means of physical activity monitoring via "Behavioural Regulation in Exercise Questionnaire"
Physical activity: questionnaire 2 | change from baseline to 12 weeks
  by means of physical activity monitoring via "Modified Baecke questionnaire"
Lung function | change from baseline to 12 weeks
  by means of general pulmonary function (spirometry, long volumes, diffusion capacity for carbon monoxide).
Heart function | change from baseline to 12 weeks
  by means of resting ECG testing

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Spruit, prof. dr., Principal Investigator — Hasselt University; Jana De Brandt, drs, Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis (ReGo), Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Brandt J, Derave W, Vandenabeele F, Pomies P, Blancquaert L, Keytsman C, Barusso-Gruninger MS, de Lima FF, Hayot M, Spruit MA, Burtin C. Efficacy of 12 weeks oral beta-alanine supplementation in patients with chronic obstructive pulmonary disease: a double-blind, randomized, placebo-controlled trial. J Cachexia Sarcopenia Muscle. 2022 Oct;13(5):2361-2372. doi: 10.1002/jcsm.13048. Epub 2022 Aug 17. PMID 35977911